CLINICAL TRIAL: NCT01935596
Title: Comparative Study of the Effects of Two Local Anesthetics Administered Intrathecally: 0.5% Levobupivacaine and Ropivacaine 0.5%
Acronym: ROPI-LEVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI09-PR-DUPONT
Record Dates: First submitted 2012-08-23; First posted 2013-09-05 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Patients Undergoing Lower Limb Surgery
Keywords: Anesthesia; Randomized study; Lower limbs surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaïne 0,5%, (Active Comparator): intrathecal administration of 15mg of ropivacaine 0.5%.
  Interventions: Drug: ropivacaïne
- lévobupivacaïne 0,5% (Active Comparator): intrathecal administration of 15mg of levobupivacaine 0.5%
  Interventions: Drug: lévobupivacaïne

INTERVENTIONS:
Drug: ropivacaïne — spinal anesthesia.
  Arms: ropivacaïne 0,5%,
Drug: lévobupivacaïne
  Arms: lévobupivacaïne 0,5%

SUMMARY:
This is a Biomedical Research, prospective, randomized, double blind, controlled monocentric, phase IV comparison of the effects of two local anesthetics intrathecally: 0.5% levobupivacaine and ropivacaine 0.5%.

DETAILED DESCRIPTION:
Progress in the practice of anesthesia led to a safety requirement of growing in daily practice. Spinal anesthesia commonly used technique for surgery of the lower limbs, provides a triple neurological lock (sensory, motor and autonomic) of roots of the spinal cord by intrathecal injection of a local anesthetic agent, following the rules of and strict aseptic conditions.

Levobupivacaine and ropivacaine local anesthetic agents are considered less toxic and tend to replace the use of bupivacaine, reference molecule, but the plasma transition is extremely toxic to patients. However, there is currently no study comparing the benefits of levobupivacaine and ropivacaine in isobaric form injected intrathecally for trauma surgery of the lower limbs. We propose to conduct a prospective, randomized double-blind comparison of the use of these two molecules in spinal isobaric form by evaluating the time and duration of action (sensory and motor block), hemodynamic and ventilatory changes (sympathetic block), and the occurrence of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to the emergency for lower limb trauma,
* age over 18 years and below 65 years
* lower limb trauma surgery can be performed under spinal anesthesia.

Exclusion Criteria:

* Refusal of patients to participate in the study,
* Patient with cons-indication to spinal anesthesia:

  * Local anesthetic allergy agents (1/13000)
  * bleeding disorders, including pharmacological origin
  * infection at the puncture site,
  * refusal of spinal anesthesia by the patient,
* Patient trust,
* Patients whose coagulation is abnormal.
* Patients with cognitive impairment or incapacitated adult,
* Multiple trauma,
* Porphyria,
* Central preexisting neuropathy,
* A history of spinal surgery,
* Epilepsy uncontrolled by treatment,
* Hypovolemia,
* Pregnant or lactating women,
* Participation in another ongoing clinical trial,
* Patient on anticoagulant therapy,
* Patient not affiliated with a social security system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
duration of anesthesia on sensitivity | during 6h after induction
  Thermo-algesic exploration of sensitivity through the application of an ice cube

SECONDARY OUTCOMES:
Duration of anesthesia on motor block | during 6h after induction

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DUPONT, Professor, Study Director — CHU Amiens France
Locations (1):
- Hervé DUPONT, Amiens, Picardie, France

REFERENCES:
- [Result] https://www.em-consulte.com/article/998410/comparaison-de-l-efficacite-de-la-levobupivacaine-